CLINICAL TRIAL: NCT02373098
Title: Effects of Fingolimod (Gilenya®) on Cytokine and Chemokine Levels in Relapsing Remitting Multiple Sclerosis Patients
Brief Title: Fingolimod Effect on Cytokine and Chemokine Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DTR04
Record Dates: First submitted 2015-02-04; First posted 2015-02-26 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Fingolimod,cytokine,chemokine,RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Intervention Model Description: A 6-month, multicenter, prospective, interventional, single arm, open label study investigating the effects of fingolimod administered according to local label recommendations on Cytokine and Chemokine Levels in Relapsing Remitting Multiple Sclerosis Patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FTY720 (Experimental)
  Interventions: Drug: Fingolimod 0.5 mg
- Healthy volunteers (No Intervention): Healthy volunteers with no intervention or drug administered.

INTERVENTIONS:
Drug: Fingolimod 0.5 mg — 66 relapsing remitting MS (RRMS) patients were recruited. Patients who met all inclusion and none of the exclusion criteria were treated by Fingolimod 0.5 mg.
  Arms: FTY720

SUMMARY:
The main purpose of this study was to measure the serum levels of cytokines and chemokines that are known to increase during multiple sclerosis relapses.

Cytokines are a broad and loose category of small proteins that are important in cell signaling.

The second purpose of the study was to test the cytokine/chemokine changes measured in the 3rd and 6th months on the efficacy parameters.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent must be obtained before the beginning of te study
2. Nonresponder RRMS patients
3. Last relapse of the patient should be at least 2 months before study entry.
4. Last interferon or glatiramer acetate dose of the patient should be at least 1 month before study entry.

Key Exclusion Criteria:

1. Patients with secondary progressive MS.
2. Patients with known contraindications for fingolimod treatment.
3. Other coexistent autoimmune diseases
4. Pregnant or nursing (lactating) women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Mecidiyeköy, Istanbul
  - Novartis Investigative Site, Üsküdar, Istanbul
  - Novartis Investigative Site, Istanbul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 healthy controls and 66 Relapsing-remitting multiple sclerosis (RRMS) patients were enrolled in the study. The healthy volunteers had only Visit 1 (Day 0). Fingolimod 0.5 mg capsule once daily was given on the same day to RRMS patients. Patients were treated for 6 months with 2 additional visits, Visit 2 and Visit 3.
Groups:
- FTY720: Relapsing-remitting multiple sclerosis (RRMS) patients were treated with fingolimod 0.5 mg capsule od.
- Healthy Volunteers: The healthy volunteers had only Visit 1 (Day 0) and served as control group for cytokine/chemokine measurements
Period: Overall Study
Arm/Group | FTY720 | Healthy Volunteers
Started | 66 | 60
Completed | 54 | 60
Not Completed | 12 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety set
Groups:
- Total: Total of all reporting groups
Arm/Group | FTY720 | Healthy Volunteers | Total
Number analyzed (Participants) | 66 | 60 | 126
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.75 (8.20) | 34.73 (9.62) | 35.27 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 40 | 86
  Male | 20 | 20 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Turkish | 66 | 60 | 126

OUTCOME MEASURES:

1. Primary Outcome: Baseline Serum Cytokine and Chemokine Levels of Healthy Controls and RRMS Patients - ELISA
Description: Blood samples were taken at baseline and measurements were performed before treatment of fingolimod.
Time Frame: Baseline
Population: Intent to treat
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- Healthy Controls: Healthy volunteers had only Visit 1 (day 0) when serum and whole blood samples were taken.
Arm/Group | Healthy Controls | FTY720
Number analyzed (Participants) | 60 | 66
pg/ml
  CCL5 (RANTES) | 212.26 (22.48) | 404.31 (55.189)
  IL-17A | 1.15 (0.03) | 1.06 (0.029)
  CXCL13 | 110.8 (22.3) | 139.68 (46.631)
  IL6 | 0.88 (0.324) | 66.53 (65.411)
  IL8 | 3.25 (0.47) | 3.57 (0.553)
  IL13 | 0.49 (0.331) | 0.3 (0.15)
  IL23 | 1.29 (0.552) | 3.04 (0.924)
  VLA4 | 1.17 (0.396) | 0.58 (0.201)
  CXCL10=IP-10 (CXCR3 ligand) | 16.09 (1.76) | 18.18 (2.405)
  CCL2=MCP-1 | 52.88 (4.281) | 62.89 (8.42)
  IL4 | 2.02 (0.077) | 2.36 (0.149)
  TNF alpha | 1.1 (0.195) | 1.06 (0.1)
  IL22 | 22.36 (0.581) | 22.41 (0.547)
Statistical Analysis 1: Comparison: Healthy Controls vs FTY720; CCL5=RANTES; Test type: Other; p = 0.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Healthy Controls vs FTY720; IL17A; Test type: Other; p = 0.035, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls vs FTY720; CXCL13; Test type: Other; p = 0.911, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Healthy Controls vs FTY720; IL6; Test type: Other; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Healthy Controls vs FTY720; IL8; Test type: Other; p = 0.934, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Healthy Controls vs FTY720; IL13; Test type: Other; p = 0.727, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Healthy Controls vs FTY720; IL23; Test type: Other; p = 0.179, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Healthy Controls vs FTY720; VLA4; Test type: Other; p = 0.208, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Healthy Controls vs FTY720; CXCL10=IP-10 (CXCR3 ligand); Test type: Other; p = 0.730, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Healthy Controls vs FTY720; CCL2=MCP-1; Test type: Other; p = 0.725, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Healthy Controls vs FTY720; IL4; Test type: Other; p = 0.057, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Healthy Controls vs FTY720; TNF alpha; Test type: Other; p = 0.724, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Healthy Controls vs FTY720; IL22; Test type: Other; p = 0.662, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Baseline Flow Cytometry Analyses for Blood Cytokines and Chemokines in Healthy Controls and RRMS Patients
Description: baseline peripheral blood flow cytometric analysis in study participants
Time Frame: Baseline
Population: Analysis was done in the healthy volunteers and RRMS patients.
Measure: Mean (Standard Error); unit: absolute cell count
Arm/Group | Healthy Controls | FTY720
Number analyzed (Participants) | 60 | 66
absolute cell count
  CD3 abs | 2048.14 (263.209) | 1610.94 (126.071)
  CD19 abs | 311.63 (57.592) | 327.63 (44.421)
  NK abs | 281.33 (39.106) | 623.57 (394.837)
  NKT abs | 135.86 (16.627) | 104.36 (15.080)
  Hi CD16CD56 abs | 26.64 (4.399) | 20.44 (3.506)
  CD4CD25 (CD3 gate) | 26.08 (3.159) | 27.08 (1.251)
  Hi CD4CD25 (CD3 gate) | 2.83 (0.383) | 3.33 (0.253)
Statistical Analysis 1: Comparison: Healthy Controls vs FTY720; CD3 abs; Test type: Other; p = 0.256, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Healthy Controls vs FTY720; CD19 abs; Test type: Other; p = 0.587, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls vs FTY720; NK abs; Test type: Other; p = 0.300, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Healthy Controls vs FTY720; NKT abs; Test type: Other; p = 0.096, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Healthy Controls vs FTY720; Hi CD16CD56 abs; Test type: Other; p = 0.270, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Healthy Controls vs FTY720; CD4CD25; Test type: Other; p = 0.902, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Healthy Controls vs FTY720; Hi CD4CD25; Test type: Other; p = 0.283, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Serum Cytokine and Chemokine Levels inRRMS Patients Between Visits
Description: Change of serum cytokine and chemokine levels measured by ELISA in RRMS patients treated with fingolimod between visits
Time Frame: Baseline, month 3, month 6
Population: Intent to treat
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- Visit 1: Relapsing-remitting multiple sclerosis (RRMS) patients were treated with fingolimod 0.5 mg capsule od at visit 1
- Visit 2: Relapsing-remitting multiple sclerosis (RRMS) patients were treated with fingolimod 0.5 mg capsule od at visit 2
- Visit 3: Relapsing-remitting multiple sclerosis (RRMS) patients were treated with fingolimod 0.5 mg capsule od at visit 3
Arm/Group | Visit 1 | Visit 2 | Visit 3
Number analyzed (Participants) | 66 | 66 | 66
pg/ml
  CXCL13=BLC | 139.68 (46.631) | 105.42 (20.61) | 105.86 (22.053)
  IL6 | 66.53 (65.411) | 49.98 (49.263) | 149.62 (144.622)
  IL8 | 3.57 (0.553) | 3.84 (0.482) | 4.29 (0.541)
  IL13 | 0.3 (0.15) | 0.35 (0.208) | 0.48 (0.289)
  CCL5= RANTES | 404.31 (55.189) | 384.12 (52.649) | 480.34 (63.874)
  IL23 | 3.04 (0.924) | 2.01 (0.629) | 2.15 (0.699)
  VLA4 | 0.58 (0.201) | 0.76 (0.356) | 0.82 (0.36)
  CXCL10=IP-10 (CXCR3 ligand) | 18.18 (2.405) | 18.46 (2.356) | 20.54 (3.008)
  CCL2=MCP-1 | 62.89 (8.42) | 74.38 (10.011) | 92.73 (13.626)
  IL4 | 2.36 (0.149) | 1.94 (0.099) | 2.12 (0.145)
  IL17A | 1.06 (0.029) | 1.09 (0.04) | 1.04 (0.033)
  TNF | 1.06 (0.1) | 1.26 (0.196) | 1.12 (0.139)
  IL22 | 22.41 (0.69) | 22.45 (0.843) | 22.99 (0.739)

4. Secondary Outcome: Peripheral Blood Cytokine and Chemokine Measurements in Healthy Controls and RRMS Patients
Description: Peripheral blood chemokine cytokine levels measured by flow cytometry during fingolimod treatment in healthy controls at baseline and in RRMS patients between visits
Time Frame: Baseline, Month 3, Month 6
Population: Intent to treat. Data analyzed in RRMS patients.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Healthy Controls | Visit 1 | Visit 2 | Visit 3
Number analyzed (Participants) | 60 | 66 | 66 | 66
pg/ml
  CD3 abs | 2048.14 (263.209) | 1610.94 (126.071) | 339.74 (43.44) | 314.75 (30.15)
  CD19 abs | 311.63 (57.592) | 327.63 (44.421) | 32.9 (5.347) | 26.56 (2.879)
  NK abs | 281.33 (39.106) | 623.57 (394.837) | 203.66 (30.487) | 181.97 (20.715)
  NKT abs | 135.86 (16.627) | 104.36 (15.08) | 88.45 (12.725) | 88.98 (11.046)
  Hi CD16CD56 abs | 26.64 (4.399) | 20.44 (3.506) | 29.35 (8.73) | 30.04 (6.59)
  CD4CD25 (CD3 gate) | 26.08 (3.159) | 27.03 (1.251) | 9.24 (1.407) | 9.22 (1.399)
  Hi CD4CD25 (CD3 gate) | 2.83 (0.383) | 3.33 (0.253) | 2.03 (0.302) | 1.77 (0.267)

5. Primary Outcome: Percent Blood Cytokines and Chemokines Via Flow Cytometry Analyses of Healthy Controls and RRMS Patients at Baseline
Description: Baseline peripheral blood flow cytometric analyses in study participants evaluated by flow cytometry analysis.
Time Frame: Baseline
Population: Analysis was done in the healthy volunteers and RRMS patients.
Measure: Mean (Standard Error); unit: Percent of cells
Arm/Group | Healthy Controls | FTY720
Number analyzed (Participants) | 60 | 66
Percent of cells
  CD3 % | 76.52 (1.494) | 71.92 (1.134)
  CD19 % | 11.57 (1.018) | 13.72 (1.336)
  NK % | 11.04 (1.328) | 10.17 (1.169)
  NKT % | 5.65 (0.855) | 5.19 (0.766)
  Hi CD16CD56 % | 1.05 (0.183) | 0.93 (0.145)
  CD3CD4 % (Lymphogate) | 41.19 (2.483) | 44.91 (1.321)
  CD3CD8 % (Lymphogate) | 23.23 (2.175) | 22.91 (1.188)
  CD3CD4 % (CD3 gate) | 57.38 (2.722) | 62.99 (1.446)
  CD3CD8 % (CD3 gate) | 35.11 (2.305) | 31.20 (1.351)
  CD4+IFNg+ (in CD4+) | 7.42 (1.994) | 3.61 (1.037)
  CD4+IL17+ (in CD4+) | 1.23 (0.173) | 1.27 (0.298)
  CD8+IFNg+ (in CD8+) | 16.45 (3.896) | 5.47 (2.463)
  CD8+IL17+ (in CD8+) | 1.71 (0.636) | 4.20 (0.923)
  IFNg+ (in CD4+CD25+) | 7.1 (1.896) | 1.98 (0.469)
  IL17+ (in CD4+CD25+) | 2.35 (0.264) | 2.06 (0.410)
  CD4+IL10+ (in CD4+) | 1.64 (0.33) | 0.72 (0.196)
  CD4+IL4+ (in CD4+) | 1.44 (0.294) | 0.96 (0.410)
  CD4-CD8-IL4+ (in CD4-CD8-) | 1.31 (0.31) | 2.62 (1.125)
  CD8+IL10+ (in CD8+) | 0.52 (0.089) | 0.31 (0.096)
  CD8+IL4+ % (in CD8+) | 5.64 (3.74) | 1.87 (0.538)
  IL10+ (in CD4+CD25+) | 2.57 (0.228) | 1.81 (0.464)
  IL4+ (in CD4+CD25+) | 1.88 (0.34) | 0.50 (0.105)
  CD4+TNFa+ (in CD4+) | 46.86 (4.892) | 23.72 (4.707)
  CD4+IL9+ (in CD4+) | 0.22 (0.109) | 0.54 (0.163)
  CD8+TNFa+ (in CD8+) | 35 (4.876) | 11.78 (2.679)
  CD8+IL9+ (in CD8+) | 0.14 (0.087) | 0.90 (0.245)
  TNFa+ (in CD4+CD25+) | 52.82 (5.019) | 23.29 (4.430)
  IL9+ (in CD4+CD25+) | 5.06 (4.497) | 0.59 (0.221)
Statistical Analysis 1: Comparison: Healthy Controls vs FTY720; CD3 %; Test type: Other; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Healthy Controls vs FTY720; CD19 %; Test type: Other; p = 0.300, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls vs FTY720; NK %; Test type: Other; p = 0.657, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Healthy Controls vs FTY720; NKT %; Test type: Other; p = 0.439, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Healthy Controls vs FTY720; Hi CD16CD56 %; Test type: Other; p = 0.449, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Healthy Controls vs FTY720; CD3CD4; Test type: Other; p = 0.356, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Healthy Controls vs FTY720; CD3CD8; Test type: Other; p = 0.787, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Healthy Controls vs FTY720; CD3CD4; Test type: Other; p = 0.121, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Healthy Controls vs FTY720; CD3CD8; Test type: Other; p = 0.209, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Healthy Controls vs FTY720; CD4+IFNg+ (in CD4+); Test type: Other; p = 0.069, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Healthy Controls vs FTY720; CD4+IL17+ (in CD4+); Test type: Other; p = 0.402, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Healthy Controls vs FTY720; CD8+IFNg+ (in CD8+); Test type: Other; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Healthy Controls vs FTY720; CD8+IL17+ (in CD8+); Test type: Other; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Healthy Controls vs FTY720; IFNg+ (in CD4+CD25+); Test type: Other; p = 0.026, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Healthy Controls vs FTY720; IL17+ (in CD4+CD25+); Test type: Other; p = 0.168, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Healthy Controls vs FTY720; CD4+IL10+ (in CD4+); Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Healthy Controls vs FTY720; CD4+IL4+ (in CD4+); Test type: Other; p = 0.013, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Healthy Controls vs FTY720; CD4-CD8-IL4+ (in CD4-CD8-); Test type: Other; p = 0.171, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Healthy Controls vs FTY720; CD8+IL10+ (in CD8+); Test type: Other; p = 0.013, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Healthy Controls vs FTY720; CD8+IL4+ (in CD8+); Test type: Other; p = 0.013, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Healthy Controls vs FTY720; IL10+ (in CD4+CD25+); Test type: Other; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Healthy Controls vs FTY720; IL4+ (in CD4+CD25+); Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Healthy Controls vs FTY720; CD4+TNFa+ (in CD4+); Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Healthy Controls vs FTY720; CD4+IL9+ (in CD4+); Test type: Other; p = 0.107, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Healthy Controls vs FTY720; CD8+TNFa+ (in CD8+); Test type: Other; p = 0.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Healthy Controls vs FTY720; CD8+IL9+ (in CD8+); Test type: Other; p = 0.022, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Healthy Controls vs FTY720; TNFa+ (in CD4+CD25+); Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Healthy Controls vs FTY720; IL9+ (in CD4+CD25+); Test type: Other; p = 0.127, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Absolute Peripheral Blood Cytokine and Chemokine Measurements in Healthy Controls and RRMS Patients
Description: Peripheral blood chemokine cytokine levels measured by flow cytometry at baseline and between visits during fingolimod treatment.
  Absolute counts of the cells were calculated according to the absolute lymphocyte counts and the percentages of cells. This allowed for a clear determination of cell counts and thus increased the reliability of the results.
Time Frame: Baseline, Month 3, Month 6
Population: Intent to treat. Data analyzed in RRMS patients.
Measure: Mean (Standard Error); unit: absolute cell count
Arm/Group | Healthy Controls | Visit 1 | Visit 2 | Visit 3
Number analyzed (Participants) | 60 | 66 | 66 | 66
absolute cell count
  CD3CD4 (Lymphogate) | 41.19 (2.483) | 44.91 (1.321) | 13.64 (1.712) | 13.9 (1.522)
  CD3CD8 (Lymphogate) | 23.23 (2.175) | 22.91 (1.188) | 32.93 (1.967) | 32.22 (2.169)
  CD3CD4 (CD3 gate) | 57.38 (2.722) | 62.99 (1.446) | 23.26 (2.726) | 24 (2.788)
  CD3CD8 (CD3 gate) | 35.11 (2.305) | 31.2 (1.351) | 59.52 (2.534) | 59.66 (2.642)
  CD4+IFNg+ (in CD4+) | 7.42 (1.994) | 3.61 (1.037) | 7.85 (2.197) | 13.97 (2.972)
  CD4+IL17+ (in CD4+) | 1.23 (0.173) | 1.27 (0.298) | 1.26 (0.224) | 2.02 (0.342)
  CD8+IFNg+ (in CD8+) | 16.45 (3.896) | 5.47 (2.463) | 5.73 (1.968) | 14.7 (3.834)
  CD8+IL17+ (in CD8+) | 1.71 (0.636) | 4.2 (0.923) | 9.22 (3.105) | 2.23 (0.505)
  IFNg+ (in CD4+CD25+) | 7.1 (1.896) | 1.98 (0.469) | 7.07 (1.719) | 9.31 (1.699)
  IL17+ (in CD4+CD25+) | 2.35 (0.264) | 2.06 (0.41) | 1.85 (0.31) | 2.7 (0.451)
  CD4+IL10+ (in CD4+) | 1.64 (0.33) | 0.72 (0.196) | 1.51 (0.422) | 2.14 (0.486)
  CD4+IL4+ (in CD4+) | 1.44 (2.94) | 0.96 (0.41) | 1.45 (0.294) | 2.32 (0.43)
  CD4-CD8-IL4+ (in CD4-CD8-) | 1.31 (0.31) | 2.62 (1.125) | 1.77 (0.267) | 2.64 (0.909)
  CD8+IL10+ (in CD8+) | 0.52 (0.089) | 0.31 (0.096) | 0.25 (0.107) | 0.67 (0.169)
  IL10+ (in CD4+CD25+) | 2.57 (0.228) | 1.81 (0.464) | 2.88 (0.471) | 4.03 (0.793)
  IL4+ (in CD4+CD25+) | 1.88 (0.34) | 0.5 (0.105) | 1.22 (0.224) | 1.49 (0.316)
  CD4+TNFa+ (in CD4+) | 46.86 (4.892) | 23.72 (4.707) | 29.45 (5.681) | 49.96 (5.832)
  CD4+IL9+ (in CD4+) | 0.22 (0.109) | 0.54 (0.163) | 0.4 (0.098) | 0.47 (0.143)
  CD8+TNFa+ (in CD8+) | 35 (4.876) | 11.78 (2.679) | 20.93 (5.361) | 41.53 (6.18)
  CD8+IL9+ (in CD8+) | 0.14 (0.087) | 0.9 (0.245) | 0.13 (0.061) | 0.14 (0.068)
  TNFa+ (in CD4+CD25+) | 52.82 (0.019) | 23.29 (4.43) | 30.39 (5.391) | 40.4 (4.907)
  IL9+ (in CD4+CD25+) | 5.06 (4.497) | 0.59 (0.221) | 0.72 (0.213) | 1.3 (0.507)

7. Secondary Outcome: Percent of Peripheral Blood Cytokine and Chemokine Measurements in Healthy Controls and RRMS Patients
Description: Peripheral blood chemokine cytokine levels measured by flow cytometry in healthy controls at baseline and in RRMS patients between visits during fingolimod treatment
Time Frame: Baseline, Month 3, Month 6
Population: Intent to treat. Data analyzed in RRMS patients.
Measure: Mean (Standard Error); unit: percent of cell count
Arm/Group | Healthy Controls | Visit 1 | Visit 2 | Visit 3
Number analyzed (Participants) | 60 | 66 | 66 | 66
percent of cell count
  CD3 % | 76.52 (1.494) | 71.92 (1.134) | 57.61 (2.401) | 59.29 (2.318)
  CD19 % | 11.57 (0.018) | 13.72 (1.336) | 6.13 (0.847) | 5.14 (0.427)
  NK % | 0.427 (1.328) | 10.17 (1.169) | 34.48 (2.758) | 33.91 (2.238)
  NKT % | 5.65 (0.855) | 5.19 (0.766) | 15.55 (1.726) | 17.66 (1.985)
  Hi CD16CD56 % | 1.05 (0.183) | 0.93 (0.145) | 5.29 (1.296) | 6.20 (1.423)
  CD8+IL4+ % (in CD8+) | 5.64 (3.74) | 1.87 (0.538) | 3.13 (0.964) | 1.91 (1.225)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Visit until 30 days after Last Patient Last Visit) up to approximately 2 years.
Description: Only patients who received at least one dose of the investigational drug (N=66) were included in the data set used for safety.
Groups:
- Fingolimod 0.5 mg: Relapsing-remitting multiple sclerosis (RRMS) patients were treated with fingolimod 0.5 mg capsule od.
- All Patients: All patients in the trial
Arm/Group | Fingolimod 0.5 mg | All Patients
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 3/66 | 3/66
Other Adverse Events (participants affected / at risk) | 7/66 | 7/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=66) | All Patients (N=66)
Sinus bradycardia (Cardiac disorders) | 2 | 2
Herpes zoster (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=66) | All Patients (N=66)
Influenza (Infections and infestations) | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Muscle contractions involuntary (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02373098/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT02373098/SAP_001.pdf